CLINICAL TRIAL: NCT01249560
Title: Impact of Raltegravir on the Viral Reservoirs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: DELLAMONICA, REDPIT
Other Study IDs: 2009 A/12
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2009-12

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- raltegravir: To illustrate the cause and effect relationship between the abnormalities of the distribution(casting) of the molecules of co-activation and the rate of apoptose, we compare also 2 groups: a first group of patients with a rate of apoptose normal ( n=10 ), and another group of patients having a rate of apoptose aggravated ( n=10 ).
  20 eligible patients will receive their treatment to J1 and will be estimated for the residual concentration of the raltegravir ®, the antiretroviral activity, the tolerance and the observance at the treatments of the study in the visits of evaluation of M1, M2, M3, M6, M12, and / or in case of premature stop(ruling) of the try(essay). Every visit will give rise to a clinical evaluation of the patient. The arisen of unwanted events

SUMMARY:
The objective of the antiretroviral treatment is to inhibit the viral replication, estimated(appreciated) by the measure of the viral plasmatic load(responsibility). In this inhibition of the viral replication usually joins an immune reconstruction [ 1 ]. Nevertheless, a viro-immunological dissociation, i.e. an undetectable viral load(responsibility) and an absence of immune reconstruction, is regularly observed. It is now turned out that an undetectable viral load(responsibility) does not correspond to the total absence of viral replication and that it is possible to detect of the intracellular pro-viral DNA . Raltegravir ®, because of its mode of action(share) inhibiting the integration of the pro-viral DNA in the chromosomes of the infected cells(units) , could decrease the intracellular reservoir of monocyte-macrophages, improve the homeostasis, so optimizing the cooperation lymphocytes T - macrophages. Several experimental data suggest that the regression of the abnormalities of cellular interactions, and the rate of apoptose abnormally raised(abnormally brought up) by cells(units) T at the patients in viro-immunological dissociation, could be obtained .

This study aims at measuring the impact of Raltegravir ® on the viral reservoirs lymphocyte and monocyte, to quantify the expression of the molecules of costimulation, the source(spring) of intercellular interactions lymphocytes - monocytes, and to measure the rate of apoptose of the cells(units) T.

DETAILED DESCRIPTION:
20 patients will be included and followed over a period of 12 months

Population of the essay

Criteria of inclusion:

Patients from 18 years to 60 years HIV + treated(handled):

* Patients presenting an undetectable viral load(responsibility) for at least 6 months and no more than year, by the use of a tritherapy containing 2 NUC + 1 IP.
* Patients presenting an immunosuppression "average" with a rate of T CD4 understood between 350 and 500 cells(units) by ml.
* Patients known for a perfect observance.

Criteria of not inclusion:

* Preliminary Use of an inhibitor of the integrase
* Patients presenting an opportunist infection and\or an evolutionary cancer
* Patients benefiting from a treatment by IL-2, interferon-alpha, steroids or the other medicines known to modify the immunity.
* Pregnant Women

ELIGIBILITY:
Inclusion Criteria:

Patients from 18 years to 60 years HIV + treated(handled):

* Patients presenting an undetectable viral load(responsibility) for at least 6 months and no more than year, by the use of a tritherapy containing 2 NUC + 1 IP.
* Patients presenting an immunosuppression "average" with a rate of T CD4 understood between 350 and 500 cells(units) by ml.
* Patients known for a perfect observance.
* Exclusion Criteria:

Preliminary Use of an inhibitor of the integrase

* Patients presenting an opportunist infection and\or an evolutionary cancer
* Patients benefiting from a treatment by IL-2, interferon-alpha, steroids or the other medicines known to modify the immunity.
* Pregnant Women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: hiv +
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-01 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Measure the effect of Raltegravir ® on the intracellular reservoirs lymphocytaires and monocytaires. | 3 months
  OBJECTIVES
  Measure the effect of Raltegravir ® on the intracellular reservoirs lymphocytes and monocytes

SECONDARY OUTCOMES:
Measure the effect of Raltegravir ® on the intracellular reservoirs lymphocytes and monocytes. | 3 months
  Secondary objectives:
  Measure the quality of the interactions lymphocytes - monocytes through the expression membranaires of the molecules of cotsimulation, the measure of proliferation, apoptose and cytokines produced via an in vitro stimulation CD3-CD28. A modulation of the cellular viral reservoirs could indeed underestimate the cellular death so schedule(program) that the profile cytokinique.
  Measure the impact of Raltegravir ® at the patients presenting an undetectable viral load(responsibility) on sub-population T CD4 and T CD8.

CONTACTS AND LOCATIONS:
Overall Officials: ROGER pierre marie, med, Principal Investigator — CHU NICE
Locations (1):
- Dellamonica, Nice, Alpes Maritimes, France